CLINICAL TRIAL: NCT02758418
Title: Efficacy of an Internet-based CBT Program for Adjustment Disorders: A Randomized Controlled Trial
Brief Title: Development and Validation of an Online Treatment Program for Adjustment Disorders
Acronym: TAO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitat Jaume I (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UJaumeI
Record Dates: First submitted 2016-04-25; First posted 2016-05-02 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Online Computerized Program Group; Waiting List Control Group
Keywords: Adjustment disorders online; Psychological Treatments; Information and Communication Technologies; Internet
MeSH Terms: interventions — Troleandomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Online Computerized Program group. (Experimental): Intervention group that uses "TAO" program.
  Interventions: Other: TAO
- Waiting list control group. (No Intervention): Participants of this group are able to access the treatment program after 7 weeks of waiting period. After this waiting period of 7 weeks, those participants still interested in receiving assistance are randomly assigned to one of two intervention conditions (Online Computerized Program group or Bibliotherapy group).

INTERVENTIONS:
Other: TAO — "TAO" is a self-applied online treatment program and consists on the computerized version of the traditional CBT protocol for Adjustment Disorders.
  The treatment protocol comprises different therapeutic components (see section Intervention) which are presented to the patients through 7 modules (one of them introductory). The Internet platform allows audiovisual resources (videos, illustrations, music and exercises that provide quick feedback) to be included, that makes the program more interactive.
  Other Names: TAO: Adjustment Disorders Online; Online Computerized CBT for Adjustment Disorders; Internet-based CBT for Adjustment Disorders
  Arms: Online Computerized Program group.

SUMMARY:
The purpose of this study is to determine the efficacy and effectiveness of a self-help treatment for adjustment disorders administered through a computerized program applied over the Internet. This treatment modality will be compared with a waiting list control group.

It is expected that, on the one side, the intervention group will improve significantly compared to the waiting list control group. On the other side, it is expected the self-applied online treatment program to be well accepted and valued by the patient.

DETAILED DESCRIPTION:
Adjustment Disorder (AD) is a highly prevalent health problem that causes a great suffering and can result in suicidal thinking and/or behavior. However, unlike mood and anxiety disorders, AD has received little attention from scientific community and very few studies have been carried out to develop evidence-based treatments (EBT) for this problem. Besides, although a cognitive behavioral therapy (CBT) protocol is currently available for the treatment of AD, many patients with this diagnosis remain untreated. There is therefore an evident need to design strategies that guarantee the patients receive adequate treatment. A feasible solution might be self-administered computerized CBT (cCBT).

A growing body of research has found that cCBT is highly effective for anxiety and depressive disorders, achieving clinical improvements similar to those obtained with traditional face-to-face interventions. The use of internet to administer EBT allows reducing the contact time between the patient and the therapist and this way reach people who otherwise would not receive treatment. Therefore, the development of a cCBT for AD will mean an improvement in the delivery and dissemination of the current treatment programs. This is especially relevant for this problem considering the scarce attention received by the scientific community and the high interference caused in the patients' life. As far as we know, there is no cCBT program specifically designed for the treatment of AD. As a consequence, further research in this area is needed.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 65 years of age.
* Meet DSM-V (APA, 2013) criteria for Adjustment Disorder.
* Be able to understand and read Spanish.
* Be able to use a computer and have an Internet connection at home.
* Have an e-mail address.
* If having any medication, not change the drug or the dose during the treatment period.

Exclusion Criteria:

* Be receiving other psychological treatment.
* Meet criteria for other severe mental disorder on Axis I: abuse or dependence of alcohol or other substances, psychotic disorder, dementia or bipolar disorder.
* Meet criteria for a severe personality disorder or illness.
* Presence of risk of suicide or self-destructive behaviors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory - Second Edition (BDI-II) (Beck, Steer, & Brown, 1996; validated in Spanish population by Sanz, Navarro, & Vázquez, 2003) score from pre-intervention to post-intervention and 3, 6 and 12 months follow-ups. | Up to 12 months
  BDI-II is a self-report inventory that measures characteristic attitudes and symptoms of depression. The total score is obtained adding the 21 items which constitute the instrument and can be a maximum of 63 points. The instrument has good internal consistency (Cronbach's alpha of 0.76 to 0.95) and a test-retest reliability of around 0.8.
Change in Beck Anxiety Inventory (BAI) (Beck & Steer, 1990; validated in Spanish population by Magán, Sanz, & García-Vera, 2008) score from pre-intervention to post-intervention and 3, 6 and 12 months follow-ups. | Up to 12 months
  BAI measures the severity of both physiological and cognitive symptoms of anxiety. The 21 items are rated on a 4-point Likert-type scale (from 0 to 3) and the total score, which oscillates between 0 and 63, is obtained after directly adding the score of each item. Psychometric analysis carried out so far show excellent internal consistency (Cronbach's alpha ≥ 0.85).

SECONDARY OUTCOMES:
Change in Inventory of Stress and Loss (Mor, Molés, Rachyla, & Quero, 2015) score from pre-intervention to post-intervention and 3, 6 and 12 months follow-ups. | Up to 12 months
  This inventory is an adaptation of the Complicated Grief Inventory (CGI; Prigerson et al., 1995). It consists of 17 first-person statements regarding the degree to which the lost person/situation interferes in the individual's life. There are 5 response options, ranging from 0 ("Never") to 4 ("Always"). The instrument has excellent internal consistency (Cronbach's alpha .86) and a test-retest reliability of around 0.90
Change in Posttraumatic Growth Inventory (PTGI) (Tedeschi & Calhoun, 1996) score from pre-intervention to post-intervention and 3, 6 and 12 months follow-ups. | Up to 12 months
  PTGI is a 21-item instrument which assesses positive outcomes reported by persons who have experienced traumatic events. A 6-point Likert response format is used, so that each statement is rated from "I did not experience this change as a result of my crisis" (scored 0), to "I experienced this change to a very great degree as a result of my crisis" (scored 5). The instrument has an excellent internal consistency (Cronbach's alpha of 0.90) and acceptable test-retest reliability of around 0.71.

OTHER OUTCOMES:
Change in Positive and Negative Affect Scale (PANAS) (Watson, Clark, & Tellegen, 1988) score from pre-intervention to post-intervention and 3, 6 and 12 months follow-ups. | Up to 12 months
  The PANAS consists of 20 items that evaluate two independent dimensions: positive affect (PA) and negative affect (NA). The range for each scale (10 items on each) is from 10 to 50. The Spanish version has demonstrated high internal consistency (0.89 to 0.91 for PA and NA, respectively, in women, and 0.87 and 0.89 for PA and NA, respectively, in men) in college students.
Change in Environmental Reward Observation Scale (EROS) (Armento & Hopko, 2007; adapted and translated into Spanish by Barraca & Pérez-Álvarez, 2010) score from pre-intervention to post-intervention and 3, 6 and 12 months follow-ups. | Up to 12 months
  EROS is a brief self-report measure of environmental reward. It consists of 10 items which are rated on a 4-point Likert-type scale. The original scale presents a good internal consistency (Cronbach's alpha of 0.85) and also a good test-retest reliability (r=0.85). The Spanish version shows similar indexes.
Change in Multidimensional Quality of Life Questionnaire (MQLI) (Mezzich et al., 1999) score from pre-intervention to post-intervention and 3, 6 and 12 months follow-ups. | Up to 12 months
  It's a 10-item self-report tool which assesses physical and emotional well-being, self-care, occupational and interpersonal functioning, community and services support, personal and spiritual fulfillment and the global perception of quality of life. The satisfaction in each of these areas is measured using a 10-point Likert rating scale. MQLI is brief and easy to administer. It also presents good internal consistency (Cronbach's alpha of 0.79) and test-retest reliability index of 0.89.
Change in Expectations and Treatment Opinion Scale (adapted from Borkovec & Nau, 1972) score from pre-intervention to post-intervention and 3, 6 and 12 months follow-ups. | Up to 12 months
  This self-report inventory measures patients' expectations before they start the treatment and their satisfaction when they complete the treatment. The 6 items are rated from 1 ("Not at all") to 10 ("Highly") and provide information about the extent to which: 1) the treatment is perceived as logic; 2) patients are satisfied with the treatment; 3) the treatment would be recommended to a friend with the same problem; 4) the treatment would be useful to treat other psychological problems; 5) patients perceive the treatment as useful for their particular problem; and 6) the treatment is perceived as aversive.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Jaume I, Castellon, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baños RM, Guillén V, Quero S, García-Palacios A, Alcañiz M, Botella C. A virtual reality system for the treatment of stress-related disorders: A preliminary analysis of efficacy compared to a standard cognitive behavioral program. Int J Hum Comput Stud 69: 602-13, 2011.
- [Background] Botella C, Baños RM, Guillén V. Una propuesta de tratamiento para los trastornos adaptativos: Creciendo en la adversidad. In: Vázquez C, Hervás G, eds. Psicología Positiva aplicada. Bilbao: Desclée de Brouwer; 2008: 129-154.
- [Background] Quero S, Andreu-Mateu S, Baños RM, Guillén V, Molés M, Botella C. Eficacia de un protocolo de tratamiento apoyado con realidad virtual para el tratamiento de los trastornos adaptativos: Un estudio controlado. Paper presented at: I Congreso Nacional de Psicología Positiva; March, 2012; Madrid, Spain.
- [Background] Quero S, Andreu-Mateu S, Moragrega I, Baños RM, Molés M, Nebot S, Botella C. Un programa cognitivo-conductual que utiliza la realidad virtual para el tratamiento de los trastornos adaptativos: Una serie de casos. Revista Argentina de Psicología Clínica. In press.
- [Background] Quero S, Moles M, Perez-Ara MA, Botella C, Banos RM. An online emotional regulation system to deliver homework assignments for treating adjustment disorders. Stud Health Technol Inform. 2012;181:273-7. PMID 22954870
- [Background] Rachyla I, Quero S, Botella C. Un tratamiento auto-aplicado a través de Internet para los Trastornos Adaptativos: Descripción de un ensayo clínico controlado aleatorizado. Paper presented at: IX Congreso de la Asociación Española de Psicología Clínica y Psicopatología (AEPCP); October, 2015; Valencia, Spain.
- [Background] Molés M. Eficacia diferencial de dos formas de aplicación de las tareas para casa en el tratamiento de los Trastornos Adaptativos: Aplicación apoyada por las TICs versus aplicación de forma tradicional [dissertation]. Castellón de la Plana, Spain: Universitat Jaume I; 2016.
- [Derived] Rachyla I, Perez-Ara M, Moles M, Campos D, Mira A, Botella C, Quero S. An internet-based intervention for adjustment disorder (TAO): study protocol for a randomized controlled trial. BMC Psychiatry. 2018 May 31;18(1):161. doi: 10.1186/s12888-018-1751-6. PMID 29855281
- See also: Psychology and Technology web platform which will include TAO (Adjustment Disorders Online), an online computerized program for the treatment of Adjustment Disorders. — http://www.psicologiaytecnologia.com/
- See also: Laboratory of Psychology and Technology of the Universitat Jaume I. — http://www.labpsitec.uji.es/eng/index.php